CLINICAL TRIAL: NCT06815042
Title: The Analysis of Efficacy Factors for Autologous Platelet-Rich Plasma Therapy in the Treatment of Elbow Tendinopathy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: CHA University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bundang_CHA
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Elbow Tendinopathy
Keywords: Platelet Rich Plasma; Protein Array Analysis; Growth factor; Patient-Rated Tennis Elbow Evaluation
MeSH Terms: conditions — Elbow Tendinopathy | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRP Treatment Arm (Experimental): Participants in this arm will receive autologous platelet-rich plasma (PRP) therapy for the treatment of elbow tendinopathy. The PRP is prepared from the patient's own blood and injected into the affected area to evaluate its clinical effectiveness. The study aims to analyze the relationship between PRP composition, including platelet concentration, white blood cell count, and specific growth factors, and treatment outcomes.
  Interventions: Biological: Autologous Platelet-Rich Plasma (PRP) Injection

INTERVENTIONS:
Biological: Autologous Platelet-Rich Plasma (PRP) Injection — Participants will receive autologous PRP injections prepared from their own blood to treat elbow tendinopathy. PRP is a plasma product with a 3-5 times higher platelet concentration than normal blood, containing growth factors such as TGF-β, PDGF, IGF, and EGF, which are known to promote tissue repair and regeneration. The PRP will be injected directly into the affected tendon area to evaluate its clinical effectiveness and the relationship between platelet concentration, growth factors, and treatment outcomes.

SUMMARY:
To identify key factors influencing the effectiveness of platelet-rich plasma (PRP) therapy in treating elbow tendinopathy, a common degenerative condition.

DETAILED DESCRIPTION:
This study focuses on evaluating the effectiveness and limitations of platelet-rich plasma (PRP) therapy in treating elbow tendinopathy, a degenerative condition that includes lateral epicondylitis (tennis elbow) and medial epicondylitis (golfer's elbow). These conditions cause pain and reduced function in the elbow, with lateral epicondylitis being more common.

PRP, a regenerative treatment made from the patient's own blood, contains platelets concentrated 3-5 times higher than normal blood, releasing growth factors like TGF-β, PDGF, IGF, and EGF, which help tissue repair. PRP therapy was first introduced for elbow tendinopathy in 2006 and has since been recognized for its potential in pain relief and healing, becoming a reimbursable treatment in Korea since 2023.

However, inconsistent clinical outcomes have been reported due to differences in PRP preparation methods and platelet concentrations. Research suggests that higher platelet counts and specific growth factors may enhance PRP effectiveness. The International Society on Thrombosis & Haemostasis classifies PRP based on platelet concentration, with some studies indicating that higher levels of TGF-β and IL-1β improve outcomes.

This study aims to identify the key components of PRP that influence treatment success, focusing on platelet concentration and growth factor levels. The goal is to establish optimal PRP preparation guidelines to ensure consistent and effective results for elbow tendinopathy, ultimately improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older
* Diagnosed with elbow tendinopathy
* Persistent pain despite receiving conservative treatment

Exclusion Criteria:

* Individuals with systemic infection at the time of study participation
* Patients with rheumatic diseases or inflammatory disorders
* Individuals with unstable systemic conditions affecting the cardiovascular, gastrointestinal, respiratory, or endocrine systems
* Any other cases deemed inappropriate for study participation by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Patient-Rated Tennis Elbow Evaluation (PRTEE) Score | Baseline, 1 week, 2 weeks and 4 weeks after the intervention
  The PRTEE is a validated questionnaire used to assess pain and functional disability in patients with elbow tendinopathy. It consists of 15 items divided into pain (5 items) and function (10 items). Scores range from 0 to 100, with higher scores indicating more severe pain and functional impairment. A decrease in score reflects improvement in symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Bundang CHA Medical Center, Seongnam-si, Gyeonggi-do, South Korea